CLINICAL TRIAL: NCT03917940
Title: The Effect of Omega 3 Fatty Acids on Blood Glucose, Lipids Profile, Serum Irisin and Sirtuin-1 in Type 2 Diabetic Mellitus Patients Treated With Glimepiride
Brief Title: Omega 3 Fatty Acids on Serum Irisin and Sirtuin-1 in Type 2 Diabetic Mellitus Patients Treated With Glimepiride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: omega 3 in diabetics type 2
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Patients
Keywords: Irisin; sirtuin-1; Omega 3 fatty acids
MeSH Terms: interventions — Fatty Acids, Omega-3; glimepiride

STUDY DESIGN:
Intervention Model Description: The patients will be divided into two groups: group 1 treated with (Omega - 3 and glimepiride, n=35). group 2 treated with glimepiride alone, n=35).
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 + glimepiride (Experimental): group 1: 35 patients treated with (Omega - 3 1000mg / day oral plus glimepiride 2mg or 3mg /day.
  Interventions: Dietary Supplement: Omega 3 fatty acids 1000 mg per day + glimepiride 2 mg or 3 mg oral
- Control (Placebo Comparator): group 2: 35 patients treated with glimepiride 2mg or 3mg /day.
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acids 1000 mg per day + glimepiride 2 mg or 3 mg oral — Omega 3 fatty acids 1000 mg per day oral
  Other Names: Omega three
  Arms: Omega 3 + glimepiride
Drug: Glimepiride — glimepiride 2 mg or 3 mg per day oral
  Other Names: Amaryl
  Arms: Control

SUMMARY:
study the effect of omega 3 fatty acids on blood glucose, lipids profile, serum Irisin and sirtuin-1 in type 2 diabetic mellitus patients treated with glimepiride.

DETAILED DESCRIPTION:
1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University
2. All Participants agreed to take part in this clinical study and provide informed consent.

Methodology

* The study will be conducted in 70 patients who are aged 30-60 years old with type 2 diabetes mellitus for at least 2 years. The patients will be assigned into two groups (Omega - 3/glimepiride, n=35; glimepiride, n=35).
* Serum Irisin, sirtuin-1, Hb A1C, Fasting blood sugar (FBS), Lipid profile, Fasting insulin, HOMA-IR and Atherogenic index of plasma (AIP) will be measured at the beginning and after 12 weeks of intervention.
* Anthro-pometric parameters including Weight and height to calculate body mass index will be measured at the beginning and after intervention.
* past medical history and medication history will be documented.
* Each subject in the test group will receive a total dose of 1000 mg of omega-3 fatty acids per day in the form of three capsules along with a glimepiride tablet to be taken once daily, while each subject in the other group will receive glimepiride tablet to be taken once daily for 12 weeks.
* Venous blood samples will be obtained from patients at the beginning and after 12 weeks of intervention.
* A commercially available enzyme-linked immuno-sorbent assay kits will be used for the measurement of Irisin and sirtuin-1.
* The patients will be advised not to change their usual diet, drug regimen and physical activity levels throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 70 Adult patients aged 30-60 years old with type 2 diabetes mellitus treated with glimepiride.
* glycated hemoglobin percent greater than 7%.
* body mass index between 25 and 35 kg/m2.
* Patients who are not consuming omega-3 fatty acids, supplements or any pharmaceutical products that may interact with their lipid profile.

Exclusion Criteria:

* Pregnant or lactating women.
* Have gastrointestinal disorders that interfere with the bowel function
* patients with severe hepatic, renal, inflammatory and thyroid diseases.
* insulin therapy.
* Have diabetes complications including micro and macrovascular complications.
* Alcoholics and patients with past history of drug abuse.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
serum Irisin concentration (ng/ml) | three months
  Myokines have anti- inflammatory properties
serum sirtuin-1 concentration (ng/ml) | three months
  class III protein deacetylase that is associated with aging, inflammation and CVD

SECONDARY OUTCOMES:
Fasting Blood Sugar | Three Months
  Serum Glucose (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Maged W Helmy, Ass. Prof., Study Director — Pharmacology & Toxicology department- faculty of pharmacy- Damanhour University.
Locations (1):
- Damanhour Medical National Institute, Damanhūr, El-Bahairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aghasi M, Ghazi-Zahedi S, Koohdani F, Siassi F, Nasli-Esfahani E, Keshavarz A, Qorbani M, Khoshamal H, Salari-Moghaddam A, Sotoudeh G. The effects of green cardamom supplementation on blood glucose, lipids profile, oxidative stress, sirtuin-1 and irisin in type 2 diabetic patients: a study protocol for a randomized placebo-controlled clinical trial. BMC Complement Altern Med. 2018 Jan 17;18(1):18. doi: 10.1186/s12906-017-2068-6. PMID 29343256
- [Result] Lluis L, Taltavull N, Munoz-Cortes M, Sanchez-Martos V, Romeu M, Giralt M, Molinar-Toribio E, Torres JL, Perez-Jimenez J, Pazos M, Mendez L, Gallardo JM, Medina I, Nogues MR. Protective effect of the omega-3 polyunsaturated fatty acids: Eicosapentaenoic acid/Docosahexaenoic acid 1:1 ratio on cardiovascular disease risk markers in rats. Lipids Health Dis. 2013 Oct 1;12:140. doi: 10.1186/1476-511X-12-140. PMID 24083393
- [Derived] Werida RH, Ramzy A, Ebrahim YN, Helmy MW. Effect of coadministration of omega-3 fatty acids with glimepiride on glycemic control, lipid profile, irisin, and sirtuin-1 in type 2 diabetes mellitus patients: a randomized controlled trial. BMC Endocr Disord. 2023 Nov 25;23(1):259. doi: 10.1186/s12902-023-01511-2. PMID 38001474